CLINICAL TRIAL: NCT07406633
Title: A Phase 2, Multicenter, Study Evaluating the Efficacy, Safety, Tolerability, Pharmacokinetics of KQB198 in Combination With Imatinib in Participants With Advanced/Metastatic GI Stromal Tumor in 1st Line Setting
Brief Title: KQB198 in Combination With Imatinib in Participants With Advanced/Metastatic GIST in 1st Line Setting
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kumquat Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KQB198-103
Record Dates: First submitted 2026-01-23; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: GIST - Gastrointestinal Stromal Tumor; GIST; GIST Metastatic Cancer; Gastro Intestinal Stromal Tumour; Gastrointestinal Tumors
Keywords: KQB198; imatinib; gleevec; gist; gastrointestinal stromal tumor; gastro intestinal stromal tumor; gist first line; gist 1st line
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Digestive System Neoplasms | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- KQB198 in Combination with Imatinib (Experimental)
  Interventions: Drug: KQB198; Drug: Imatinib (Gleevec)

INTERVENTIONS:
Drug: KQB198 — Oral KQB198
Drug: Imatinib (Gleevec) — Oral Imatinib

SUMMARY:
This study will test an experimental drug called KQB198 in combination with imatinib. The goal is to determine if this combination is safe and tolerable and assess how effective the combination is at treating GIST. Imatinib has been approved by the FDA for the treatment of different types of cancer including GIST.

ELIGIBILITY:
Inclusion Criteria

All Participants:

* Unresectable or metastatic disease
* Tissue confirmation of GIST
* Valid results from local testing of blood or tumor tissue documenting the presence of a KIT mutation (must not have exon 9 mutation) or PDGFRA mutation (must not have PDGFRA D842V).
* Measurable disease per RECIST v1.1.
* Patients must be in 1st line of treatment for advanced or metastatic disease. Prior imatinib is allowed in adjuvant or neoadjuvant setting, as long as imatinib was stopped over 1 year ago.
* Adequate organ function and performance status

Exclusion Criteria

Participants are excluded from the study if any of the following criteria apply:

* Unable to swallow or GI condition that prevents absorption.
* Other active malignancies within the last 2 years.
* History of hypersensitivity to any component of KQB198 or imatinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 30 months
  Evaluate efficacy of study treatment, as measured by Objective Response Rate (ORR) using Response Evaluation Criteria in Gastrointestinal Stromal Tumors (GIST). Objective response is the proportion of subjects that experience confirmed complete response (CR) or partial response (PR) based on RECIST v1.1 during the time period from 1st dose of study treatment until last dose.

SECONDARY OUTCOMES:
Duration of response (DOR) | 30 months
  Duration of response defined as the time from date of the first documentation of objective tumor response (CR or PR) based on RECIST v1.1 to the first documentation of either PD or death due to any cause, whichever occurs first.
Disease control rate (DCR) | 30 months
  Disease control rate is the proportion of subjects that experience confirmed complete response (CR), partial response (PR), or stable disease based on RECIST v1.1 during the time period from 1st dose of study treatment until last dose.
Time to response (TTR) | 30 months
  Time to response is defined as time from 1st dose of study treatment to date of 1st documentation of objective tumor response (CR or PR) based on RECIST v1.1.
Progression-free survival (PFS) | Up to 30 months
  Progression-free survival is defined as the time from enrollment to the date of Progressive Disease (PD) based on RECIST v1.1 or death due to any cause, whichever occurs first. PFS at 6 months will also be characterized which indicates the proportion of subjects that experience progression within 6 months from time of enrollment.
Overall survival (OS) | Up to 30 months
  Evaluate efficacy of study treatment characterized by OS. Overall survival is defined as the time from start of treatment to death.
Number of patients who experience treatment-emergent adverse advents, serious adverse events, and dose-limiting toxicities (Part 1) | From enrollment to the end of treatment
  Safety characterized by type, incidence, severity, timing, seriousness and relationship to study treatment of adverse events (AEs), serious adverse events (SAEs), and dose limiting toxicities (DLTs), from first dose of study treatment to 28 days after last dose of study treatment.
Area under the curve (AUC) | Up to 30 months
  Area under the concentration-time curve (AUC) of KQB198 in combination with imatinib.
Maximum plasma concentration (Cmax) | Up to 30 months
  Maximum plasma concentration (Cmax) of KQB198 in combination with imatinib.
Time to maximum plasma concentration (Tmax) | Up to 30 months
  Time to maximum plasma concentration (Tmax) of KQB198 in combination with imatinib.

IPD SHARING:
Plan to Share IPD: No